CLINICAL TRIAL: NCT04168398
Title: Clopidogrel Aspirin Therapy (CAT) Versus Apixiban Aspirin Therapy (AAT) After Lower Limb Revascularization
Acronym: CVAALR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nshaat Elsaadany, Principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R.19.06.544.R1 - 2019/07/03
Record Dates: First submitted 2019-10-25; First posted 2019-11-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Ischemia; Anticoagulants
Keywords: Clopidogrel, Apixiban and Lower Limb Revascularization
MeSH Terms: conditions — Ischemia | interventions — Drug Combinations

STUDY DESIGN:
Intervention Model Description: Randomized controlled Prospective study: It will include all patients presented to our department fulfilling the inclusion criteria. We revascularize about 5-10 limbs per week and the study will be carried over 30 months; sample size will be 600-1200 patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Block randomization: Two elements A for CAT, B for AAT A A B B A B A B A B B A B B A A B A B A B A A B
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Plavix 75mg and juspirin 81 mg therapy (Experimental): Clopidogrel 75 mg (Plavix 75mg) plus Aspirin (juspirin) 81 mg.
  Interventions: Drug: Combination drug
- Eliquis 2.5mg and juspirin 81 mg therapy): (Experimental): Apixiban 2.5 twice daily (Eliquis 2.5mg) plus Aspirin (juspirin) 81 mg.
  Interventions: Drug: Combination drug

INTERVENTIONS:
Drug: Combination drug — Anticoagulation
  Other Names: anticoagulations plus antiplatelets

SUMMARY:
the Aim of the work is to compare the effect of CAT (Clopidogrel aspirin therapy) and AAT (Apixiban aspirin therapy) after lower extremity revascularization.

The study will be conducted at the department of vascular surgery in Mansoura university hospitals in a randomized controlled Prospective study over 2 years: 2019-2021. It will include all patients presented to our department fulfilling the ,We revascularize about 5-10 limbs per week and the study will be carried over 30 months; sample size will be 600-1200 patients,The study will be conducted in patients with lower limb ischemia who need revascularization. All Symptomatic peripheral artery disease according to Rutherford stages 3 to 6; will be included Patients with severe groin or limb infection, can't give consent (unconscious) and those with mental or behavioral disorders; will be excluded.

Therapies:CAT (Clopidogrel aspirin therapy) Clopidogrel 75 mg (Plavix 75mg) plus Aspirin 81 mg. AAT (Apixiban aspirin therapy): Apixiban 2.5 twice daily (Eliquis 2.5mg) plus Aspirin 81 mg. Every patient will be followed every week till first month, then every 3 months till 1 years. Hemodynamic improvement was assessed by ankle brachial pressure index (ABI), performed before and after the procedure and every 3 months. Evaluation made by CTA or duplex ultrasonography to determine 1ry and 2ry patency, Coagulation profile (platelet count, INR, prothrombin time and activated partial thromboplastin time). Adverse bleeding complications will be documented

DETAILED DESCRIPTION:
INTRODUCTION:

Atherothrombotic disorders of the cerebrovascular, coronary, and peripheral arterial circulation, affect nearly 20-30% of those older than 70 years of age and are among the leading causes of death and disability in the world. Individuals with peripheral artery disease (PAD), referring to arterial vascular disease of the extremities, have the greatest risk of experiencing cardiovascular death and myocardial infarction when compared to those with coronary artery disease or cerebrovascular disease alone PAD usually signals more systemic atherosclerotic disease and often goes undiagnosed and undertreated, which is thought to be a major reason for why these patients have been found to be at increased risk for major adverse cardiovascular events and mortality. One of the major goals of antiplatelet therapy is for prevention, both primary and secondary, of acute thrombotic events. Despite the increased local and systemic cardiovascular risk in PAD patients, the literature on the most effective antiplatelet regimen and its recommended duration are lacking, especially compared to studies primarily focusing on coronary artery disease. The major consensus guidelines for PAD suggest using mono antiplatelet therapy in PAD but state that the data either for or against the use of DAPT in this population are too limited to make strong recommendations. There has been an attempt to update the international TASC guidelines but disagreement among the societies has delayed a universally accepted TASC III document. After PAD revascularization, corresponding risks are even higher, with reported rates of nonfatal MI, ischemic stroke, or cardiovascular death 36 months after procedure of 14% among patients with IC and 34% among those with CLI. These risks are further elevated after repeat limb revascularization, supporting the need for more aggressive secondary prevention measures, including intensive antithrombotic therapy, to prevent recurrent events in this high-risk population. Despite the greater risk of cardiovascular and limb adverse outcomes in patients with PAD undergoing limb revascularization, high-quality data on antithrombotic therapy in this clinical context are sparse. As a result, recommendations regarding antithrombotic therapy for these patients are based on lower levels of evidence and are inconsistent.

Until now no clinical trial had reported the use of AAT (Apixiban aspirin therapy) after lower limb revascularization therefore, the purpose of this study is to evaluate and compare the effect of CAT (Clopidogrel aspirin therapy) and AAT (Apixiban aspirin therapy) at time of discharge, on survival following lower extremity revascularization and major adverse effects Aim of the work compare the effect of CAT (Clopidogrel aspirin therapy) and AAT (Apixiban aspirin therapy) after lower extremity revascularization.

Outcome Primary outcomes: Major adverse limb events (MALES);

* Endovascular or surgical revascularization
* Acute vessel thrombosis,
* Amputation of the target limb Secondary outcomes: Major adverse cardiovascular events (MACE);
* Nonfatal stroke
* Nonfatal myocardial infarction
* Cardiovascular death. Patients and methods Study location: The study will be conducted at the department of vascular surgery in Mansoura university hospitals Type of study: Randomized controlled Prospective study Study duration: 2 years: 2019-2021 Sample size: It will include all patients presented to our department fulfilling the inclusion criteria. We revascularize about 5-10 limbs per week and the study will be carried over 30 months; sample size will be 600-1200 patients Study population: The study will be conducted in patients with lower limb ischemia who need revascularization.

Inclusion criteria: Symptomatic peripheral artery disease according to Rutherford stages 3 to 6.

Exclusion criteria

1. Patients with severe groin or limb infection.
2. who can't give consent (unconscious)
3. Those with mental or behavioral disorders will be excluded. Consent: Patients after signing informed consent that possible complication from the procedure ought to happen and what are the alternatives.

Data collection: The demographics, Symptoms and preoperative clinical data will be collected History Data: included patient's demographics, underlying medical conditions, any previous associated morbidity.

Examination: Arterial assessments. Laboratory: Blood picture, Blood sugar level, Kidney functions, Liver functions and Coagulation profile.

Imaging: Duplex US and CTA Method of Randomization: Block randomization: Two elements A for CAT, B for AAT A A B B A B A B A B B A B B A A B A B A B A A B Therapies CAT (Clopidogrel aspirin therapy) Clopidogrel 75 mg (Plavix 75mg) plus Aspirin 81 mg.

AAT (Apixiban aspirin therapy):

Apixiban 2.5 twice daily (Eliquis 2.5mg) plus Aspirin 81 mg. Follow up

* Every patient will be followed every week till first month, then every 3 months till 1 years.
* Hemodynamic improvement was assessed by ankle brachial pressure index (ABI), performed before and after the procedure and every 3 months.
* Evaluation made by CTA or duplex ultrasonography to determine 1ry and 2ry patency
* Coagulation profile (platelet count, INR, prothrombin time and activated partial thromboplastin time).
* Adverse bleeding complications.
* Both MACEs and MALEs will be documented Statistical analysis
* The data will be analyzed using Statistical Package for the Social Sciences. The numerical outcomes e.g. age is calculated as mean. Gender will be recorded as frequency and percentage. Chi Square test is applied to assess the association of various parameters. The results will be considered statistically significant if the p-value is found to be less than or equal to 0.05.

ELIGIBILITY:
Inclusion Criteria:

Symptomatic peripheral artery disease according to Rutherford stages 3 to 6.

Exclusion Criteria:

1. Patients with severe groin or limb infection.
2. who can't give consent (unconscious)
3. Those with mental or behavioral disorders will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1536 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Major adverse limb events (MALES); | two year
  * Endovascular or surgical revascularization
  * Acute vessel thrombosis,
  * Amputation of the target limb

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE); | two year
  * Nonfatal stroke
  * Nonfatal myocardial infarction
  * Cardiovascular death.

CONTACTS AND LOCATIONS:
Overall Officials: Nshaat A Elsaadany, MSc, Principal Investigator — Mansoura University
Locations (1):
- Mansoura, Al Mansurah, Mansoura University, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The demographics, Symptoms and preoperative clinical data will be collected History Data: included patient's demographics, underlying medical conditions, any previous associated morbidity.
  Examination: Arterial assessments. Laboratory: Blood picture, Blood sugar level, Kidney functions, Liver functions and Coagulation profile.